CLINICAL TRIAL: NCT05029440
Title: Effect of Full-Body Pulsed Electromagnetic Field Versus Pulsed High Intensity Laser Therapy in the Treatment of Patients With Osteopenia or Osteoporosis
Brief Title: Pulsed Electromagnetic Field Versus Pulsed High Intensity Laser in the of Osteoprosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm AlQura U
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Osteopenia or Osteoporosis
Keywords: T-scores of ≤1.5
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electromagnetic and Exercise Group (Experimental): Pulsed Electromagnetic Field (PEMF) PEMF was administered to the whole body using a 1.8×0.6m mat Exercise Program Exercise program to facilitate bone health
  Interventions: Other: Pulsed Electromagnetic Field; Other: Exercise Program
- Laser and Exercise Group (Active Comparator): Pulsed High Intensity Laser Therapy (HILT) HILT was administered to lumbar region and femoral head using Exercise Program Exercise program to facilitate bone health
  Interventions: Other: Exercise Program; Other: Pulsed High Laser Therapy
- Exercise Group (Active Comparator): Exercise Program Exercise program to facilitate bone health
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Pulsed Electromagnetic Field — PEMF was administered to the whole body for PEMF groups using a 1.8×0.6m mat 30 minutes/day, 3 times/week for 3 months.
  Arms: Electromagnetic and Exercise Group
Other: Exercise Program — The exercise training program included treadmill and aerobic exercises for hip and upper limb and performed for 50 minutes.
Other: Pulsed High Laser Therapy — High Laser was delivered with a total dose of energy of 3000 J was delivered in two treatment phases. The initial phase was performed with fast manual scanning at 510, 610, and 710 mJ/cm2 in three successive subphases and 500 J in each subphase for a total of 1500 J. The final phase was the same as the initial phase except that the scanning was slow. The average area for the upper thigh or lower back was 200 cm2 with an average fluency of 15 J/cm2 and the application time for each area was 18 min. HILT was applied using a HIRO 3 device (ASA, Arcugnano, Vicenza, Italy).
  Arms: Laser and Exercise Group

SUMMARY:
Osteoporosis is the most prevalent metabolic bone disease. Although osteoporosis is widely considered to be much more prevalent in women approximately 39% of new osteoporotic fractures estimated to have occurred Worldwide in 2000 were in men. A number of studies investigate the effect of physical therapy modalities in treatment of osteoporosis. The use of pulsed electromagnetic field (PEMF) represents an attractive alternative for Osteoporosis. Previous studies suggested that pulsed electromagnetic field could be beneficial for increase bone mineral density in osteoporotic patients, but there is a lack of Knowledge about the comparison with pulsed high laser therapy.

DETAILED DESCRIPTION:
Objectives: This randomized controlled study aims to investigate theEffect of Full-Body Pulsed Electromagnetic Field versus Pulsed High Intensity Laser Therapy in the Treatment of Men with Osteopenia or Osteoporosis Methods: Ninty male patients with osteopenia or osteoporosis will participate in this study, their age ranges between 30-60 years. They have BMD T-scores ≤ - 1.5. All patients will be randomized into one of three groups. Group one received PEMF and exercise (PEMF+EX), group two received HILT and exercise (HILT+EX) and group three will be treated by exercise alone (Ex). The exercise training program will include treadmill and aerobic exercises for hip and upper limb will be performed for 50 minutes.PEMF was administered to the whole body for PEMF groups using a 1.8×0.6m mat 30 minutes/day, 3 times/week for 3 months. Dual-energy X-ray absorptiometry (DEXA) will assess Bone mineral density BMD (g/cm2), bone mineral content (BMC), T-Score and Z-Score at the lumbar spine, proximal femur and forearm region, bone markers (25-hydroxy Vit D , Total, undercarboxylated Ostocalcin, Parathyroid Hormone, Total and Ionized calcium and Alkaline Phosphatase (ALP), also will be measured. The assessment will be done at baseline, after treatment (12 weeks) and after 6 months as follow up. The data will be analyzed using repeated measures Analysis of variance (ANOVA) for comparison between pre-treatment and post treatment measurement intervals. One-way ANOVA is used to compare between each treatment interval in treatment groups at pre-test and post treatment measurement intervals. The level of significance is set at 0.05 for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a T-scores of ≤ #1.5, all patients received the same medical treatment for osteoporosis and the same average blood glucose level, sufficient ability to understand the nature and potential risks of the study.

Exclusion Criteria:

* Diabetes mellitus, ischemic heart disease, arrhythmia, uncontrolled thyroid disease, cardiac pacemaker, tuberculosis, neuropsychiatric disorders (dementia, cerebrovascular disease, alcohol abuse, severe depression, panic disorder, bipolar disorder, or psychosis), and malignancy.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline Bone Mineral Density at 3 months | Baseline and 3 months post-intervention
  Bone Mineral Density was assessed by the DEXA in the lumbar spine, proximal femur and forearm region in g/cm2.
Change from baseline Vitamin D levels at 3 months | Baseline and 3 months post-intervention
  Vitamin D test is the most accurate way to measure how much vitamin D is in the body. Vitamin D in serum was measured as a standard procedure at the Department of Clinical Chemistry.
Change from baseline Alkaline Phosphatase at 3 months | Baseline and 3 months post-intervention
  Alkaline Phosphatase was estimated colorimetric end point and kinetic using fully automated analyzer Advia Centaur, according to enclosed pamphlet.

SECONDARY OUTCOMES:
Change from baseline Osteocalcin at 3 months | Baseline and 3 months post-intervention
  Ostocalcin is a predictive marker for osteoprosis and bone fracture. Serum Osteocalcin was measured in serum samples using an ELISA Kits.
Change from baseline Parathyroid Hormone at 3 months | Baseline and 3 months post-intervention
  Parathyroid hormones (PTH) was measurement chemiluminescence immunoassays [QuiCkIntraOperativeTM intact PTH. The assay was performed on the Immuno- automated analyzer (DPC) at the Department of Clinical Chemistry at Um ALQURA University, Faculty of Applied Medical Science. The Roche intact-PTH test was assayed on an Elecsys-1010 immunoassay analyzer (Roche Diagnostics) with its "Stat-function.

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M Elshamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Al Noor Specialized Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No